CLINICAL TRIAL: NCT03517215
Title: The Development and Testing of a Scaling Strategy for a Community-based Primary Care Antimicrobial Stewardship Program Utilizing an Innovative University of Toronto Primary Care Testing Platform: the UTOPIAN Practice Based Research Network
Brief Title: The Development and Testing of a Scaling Strategy for a Community-Based Primary Care Antimicrobial Stewardship Program
Acronym: PC-ASP 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: Sinai Health System (Other)
Responsible Party: Principal Investigator, Warren McIsaac, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-0016-E
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Acute Rhinosinusitis; Sore Throat; Acute Cystitis; Acute Bronchitis
MeSH Terms: conditions — Pharyngitis; Bronchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced CB-ASP (Experimental): If a site is randomized to the enhanced CB-ASP, prescribers at that site will be required to attend an education session. In the four months following the initial session, prescribers will be asked to complete one on-line eModule for each target condition (acute sinusitis, sore throat, acute bronchitis and acute uncomplicated cystitis) each month. Each module will take approximately 15 minutes to complete. Two audit and feedback reports (every 3 months) of their clinic's prescriptions for these conditions will be provided where they will be asked to review and discuss with their colleagues and study staff.
  Interventions: Behavioral: Enhanced CB-ASP
- Standard CB-ASP (Active Comparator): If a site is randomized to the standard CB-ASP strategy arm, prescribers will be offered the opportunity to attend the 1 hour introductory seminar by a web-link, provided with access to the short e-learning modules each month by email, and sent their clinic's audit and feedback reports by email for review two times during the study.
  Interventions: Behavioral: Standard CB-ASP
- Control (No Intervention): If a site is randomized to the control arm, the site will not receive any active interventions. Prescribers at the site will be offered access to the eModules at the completion of the study and provided with one audit and feedback report of their clinic's antibiotic prescribing patterns for local quality improvement needs as desired.

INTERVENTIONS:
Behavioral: Enhanced CB-ASP — The education session will be a 1-hour on site presentation that will cover antimicrobial resistance, antimicrobial stewardship, an introduction to effective primary care interventions for reducing antibiotic prescribing, and a review of the clinic's baseline audit of antimicrobial prescribing for the prior year. E-Modules will be completed online and audit and feedback sessions will be held in person to give an overview of each clinic's prescribing numbers.
  Arms: Enhanced CB-ASP
Behavioral: Standard CB-ASP — A one hour introductory educational seminar will be offered to prescribers via a web-link. They will be provided with access to e-modules each month by email and sent their audit and feedback reports by email.
  Arms: Standard CB-ASP

SUMMARY:
Antibiotic resistant infections are expected to cause 10 million deaths worldwide by 2050, and exceed cancer deaths. Reducing antibiotic use can reduce resistance levels. Hospitals have now developed Antimicrobial Stewardship Programs that promote better use of antibiotics. However, 80% of antibiotics are prescribed in the community where stewardship programs do not exist. Antibiotics are often prescribed for coughs and colds, where it can be difficult to tell if these are cases of pneumonia or strep throat. Doctors may prescribe antibiotics 'just in case' and patients may request antibiotics hoping to feel better faster. To help family doctors and patients, a team of infectious disease specialists, researchers and community family physicians have collaboratively developed an Antimicrobial Stewardship Program (ASP) for use in the community. Testing in 3 family medicine clinics is showing reduced antibiotic use. What is needed is a strategy to 'scale' up this program province wide to reduce antibiotic use enough to reduce resistance levels, but how to do this is not known. Working with a community clinic network, this project will test two implementation strategies to inform how best to implement a Community-Based ASP.

DETAILED DESCRIPTION:
Antimicrobial resistance is evolving globally. The latest 'superbug', plasmid mediated colistin resistant E.coli (MDR-1), identified in North America highlights this. Previously, colistin was the drug of last resort that could be used for organisms resistant to all other antibiotics. Current projections are that by 2050, there will be 10 million deaths annually from antimicrobial resistant infections, and this will exceed deaths from cancer.

Antibiotic overuse is considered a main factor in promoting antimicrobial resistance. Countries with high volumes of antibiotic use have higher levels of resistant organisms. After a single antibiotic course, a person's risk of acquiring an antimicrobial resistant infection is increased. Recognizing the need for action to address this crisis, governments in the United States and Canada have issued recent policy statements calling for, among other actions, reductions in antibiotic overuse. Over 80% of antibiotics in Canada are prescribed in the community for common respiratory and other infections. Currently, this amounts to one antibiotic prescription issued for every 6 Canadians each year.

In an ongoing 2014-15 Innovation Fund grant (Community ASP-Phase 1), a team of infectious disease experts and pharmacists with hospital ASP experience, community family physicians working in primary care clinics, and researchers with expertise in community infections collaboratively developed a Community-Based Primary Care Antimicrobial Stewardship Program(CB-ASP). Preliminary results (presented below) show positive effects on key antibiotic utilization parameters. What is needed now is a strategy to 'scale' this program up to similar clinics province wide. This will be necessary to achieve the reduction in the volumes of antibiotic use needed to reduce resistance. Exactly the optimal way to do this and what resources will be needed is not known. Providing the answers to these questions are the objectives of this proposal (CB-ASP -Phase 2).

Objectives - This study will seek to determine the best way for the developed CB-ASP to be successfully scaled up to other family medicine clinics, by testing strategies that are resourced with different intensities, utilizing an innovative primary care research platform.

Study Design - This study will be a 9-month cluster randomized trial over one winter of a less resource intensive and more resource intensive scaling strategy for disseminating a Community-Based Antimicrobial Stewardship Program (CB-ASP) in 6 clinics within a network (UTOPIAN) of linked primary care practices, stratified by small verses large urban center.

This study will test different levels of support (resources provided) in delivering a clinic-based, educational, community-focused ASP intervention directed at family physicians and nurse practitioners. These health professionals are licensed to prescribe antibiotics in these settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults who present with an illness consistent with one of the following conditions, as judged by the prescriber: a sore throat presentation (either pharyngitis, tonsillitis), an uncomplicated upper respiratory infection (URI; ie- the common cold), acute sinusitis, acute bronchitis, or non-pregnant women who present with acute uncomplicated cystitis.

Exclusion Criteria:

* pregnant women or male urinary tract infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in antibiotic prescribing | 9 months
  To determine the proportion of antibiotics prescribed for pharyngitis, tonsillitis, acute sinusitis and acute bronchitis

SECONDARY OUTCOMES:
Use of delayed antibiotic prescriptions | 9 months
  Assess the proportion of delayed prescription issued during the post intervention phased compared to the before
Reduction in the duration of prescriptions | 9 months
  Assess where there was a reduction in the duration of prescriptions
Specific antibiotics prescribed | 9 months
  Assess the specific antibiotics prescribed and if there is a reduction in the use of broad spectrum antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Warren McIsaac, MD, Principal Investigator — Sinai Health System
Locations (3):
- Canada (3):
  - North York General Hospital, North York, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Granovsky Gluskin Family Medicine Cwntre, Toronto, Ontario

REFERENCES:
- [Derived] McIsaac W, Kukan S, Huszti E, Szadkowski L, O'Neill B, Virani S, Ivers N, Lall R, Toor N, Shah M, Alvi R, Bhatt A, Nakamachi Y, Morris AM. A pragmatic randomized trial of a primary care antimicrobial stewardship intervention in Ontario, Canada. BMC Fam Pract. 2021 Sep 15;22(1):185. doi: 10.1186/s12875-021-01536-3. PMID 34525972